CLINICAL TRIAL: NCT02835157
Title: Multiple Electrolyte Solution vs. Saline in Pediatric Septic Shock
Brief Title: Balanced Crystalloid vs. Saline in Children With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); St Johns Medical College Hospital, Bangalore, India (Other)
Responsible Party: Principal Investigator, Jhuma Sankar, Additional Professor Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC/NP-424/09.10.2015
Record Dates: First submitted 2016-03-01; First posted 2016-07-15 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Septic Shock; Shock
Keywords: Normal saline; Multiple electrolyte solution; Septic shock; Children; Hyperchloremia; Acute kidney injury; 0.9% saline; Balanced crystalloid
MeSH Terms: conditions — Shock, Septic; Shock; Acute Kidney Injury | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The enrolled children will be randomized to either balanced crystalloid (Plasma-Lyte A or multiple electrolyte solutions or MES group) or 0.9% saline (saline group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Serially numbered, sealed, opaque pouches containing 10 bags of 500 ml of either MES or saline each will be kept at the study site. Each of the 500 ml bags will be packed in sealed opaque covers inside the pouches as well.The research staff will pick the bag of fluids kept as per allocation sequence and start the bolus in the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced crystalloid or multiple electrolyte solution group (Experimental): After enrollment, a fluid bolus comprising of 'multiple electrolyte solution (Plasma-Lyte P)' solution at a dose of 20 ml/kg over 15-20 minutes (recommended) with careful monitoring for features of fluid overload would be administered to each child. Fluid resuscitation will be targeted at achieving the therapeutic end points as given in study definitions. After this the management protocol will be as per recommendations of the American College of Critical Care Medicine 2017 for septic shock in children.
  Interventions: Drug: Balanced crystalloid solution
- 0.9% saline or saline group (Active Comparator): After enrollment, a fluid bolus comprising of 'saline' solution at a dose of 20 ml/kg over 15-20 minutes (recommended) with careful monitoring for features of fluid overload would be administered to each child. Fluid resuscitation will be targeted at achieving the therapeutic end points as given in study definitions. After this the management protocol will be as per recommendations of the American College of Critical Care Medicine 2017 for septic shock in children.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: Balanced crystalloid solution — Multiple electrolyte solution as boluses would be administered.
  Other Names: Plasma-Lyte A 148; Multiple electrolyte solution
  Arms: Balanced crystalloid or multiple electrolyte solution group
Drug: 0.9%sodium chloride — saline as boluses would be administered
  Other Names: Saline
  Arms: 0.9% saline or saline group

SUMMARY:
Fluid resuscitation is the cornerstone of pediatric shock management; current practices of fluid resuscitation in children are not evidence based. Normal saline is the preferred crystalloid recommended during initial resuscitation in shock, as the incidence of hyponatremia is lower with normal saline compared to all other fluids available and commonly used. However, normal saline has its own set of undesired physicochemical actions. Emerging data strongly indicate the increased incidence of hyperchloremia, metabolic acidosis and consequently, acute kidney injury associated with infusion of large volumes of normal saline. Balanced salt solutions or crystalloids, which have composition resembling plasma but lower chloride concentrations than normal saline, clearly decrease the risk of hyperchloremia and metabolic acidosis in adult as well as pediatric studies when used during the peri-operative period. The results favored balanced solutions in comparison to normal saline. Recent systematic reviews comparing balanced or buffered versus non-buffered fluids for surgery in adults favored the former solution as the metabolic derangements were less with the use of this type of fluid. In adult patients, the two solutions have been compared in various other settings as well such as in traumatic brain injury and in shock. The results favored balanced solutions in comparison to normal saline. However, in the non-surgical setting there is a paucity of evidence on the use of these solutions in children with shock and more evidence needs to be generated to support or refute the use of this fluid as compared to normal saline.

Given this background, the investigators decided to compare the effect of two solutions on the incidence of acute kidney injury in children resuscitated with either of the two fluids. Children receiving at least one fluid bolus at 20 ml/kg in the first hour would be enrolled and followed up for the proposed outcome variables. The investigators plan to enroll 708 patients over a period of 3 years. The investigators believe that the proposed study will provide answer to the research question of which of the fluids could be preferred for resuscitation.

DETAILED DESCRIPTION:
Background

Fluid resuscitation is the cornerstone of pediatric shock management; current practices of fluid resuscitation in children are not evidence based. Emerging data strongly indicate the increased incidence of hyperchloremic metabolic acidosis and consequently, acute kidney injury associated with infusion of large volumes of normal saline in critically ill adults in shock. Balanced salt solutions or crystalloids, which have composition resembling plasma but lower chloride concentrations than normal saline, have shown to decrease the risk of hyperchloremia and metabolic acidosis in adult as well as pediatric studies when used during the peri-operative period. In adult patients, the two solutions have been compared in various other settings as well such as in traumatic brain injury and in shock. The results favored balanced solutions in comparison to normal saline. However, in the non-surgical setting there is a paucity of evidence on the use of these solutions in children with shock and more evidence needs to be generated to support or refute the use of this fluid as compared to normal saline.

Objectives

Primary To examine if use of 'balanced crystalloids (multiple electrolyte solution)" results in lower incidence of new or progressive Acute kidney injury (defined as increase in serum creatinine by > 0.3mg/dL within 48 hours or to 1.5 times baseline or more within the last 7 days or urine output less than 0.5 mL/kg/h for 6 hours) in the first seven days after initial fluid resuscitation as compared to saline.

Secondary

To evaluate the difference if any, between two fluid types with regard to the following secondary objectives such as:

1. Incidence of hyperchloremia (defined as serum chloride levels >108 mEq/L) at 6, 24, 48 and 72 hrs of fluid resuscitation.
2. Incidence of metabolic acidosis at 6, 24, 48 and 72 hrs of fluid resuscitation.
3. Requirement of fluid boluses in first 6 hrs and total fluids in first 24 hours, 48 hours and 72 hours.
4. Proportion of patients achieving the pre-determined therapeutic end points at 6, 24, 48 hours and 72 hours after fluid resuscitation.
5. Need for inotrope therapy in first 7 days.
6. Change in SOFA scores and PELOD scores at 24 hours and 48 hours.
7. Time to resolution of AKI.
8. In- ICU mortality rates.
9. Ventilator free days, ICU free days and Hospital free days.

Site of study

Pediatric emergency and PICU, Department of Pediatrics, All India Institute of medical Sciences,New Delhi

Other sites

PGIMER, Chandigarh, JIPMER Puducherry and St Johns Medical College Bengaluru

Study Design

Randomized controlled trial (safety and superiority for kidney injury). Multicenter trial.

Study Duration

3 years

Study definitions

Septic shock is defined as children who have a suspected infection manifested by hypothermia or hyperthermia and have at least two clinical signs of decreased perfusion with or without hypotension such as decreased mental status, prolonged capillary refill of >2 secs (cold shock) or flash capillary refill (warm shock), diminished (cold shock) or bounding (warm shock) peripheral pulses, mottled cool extremities (cold shock), or decreased urine output of <1 ml/kg/hr).

Therapeutic end points

* Normal heart rate
* Appropriate-for-age mean arterial pressure (MAP) measured non-invasively;
* Normal pulses with no difference between peripheral and central pulses, warm extremities;
* Capillary refill time <2 seconds;
* Normal mental status;
* Urine output ≥ 1mL/kg/hr,

Hyperchloremia: Defined as serum chloride value of >108 meq/L, based on our laboratory cut off of 98-108 meq/L Metabolic acidosis: pH of less than 7.35 with serum bicarbonate < 24 meq/L with low to normal pCO2 (<40 mm Hg)

Acute kidney injury: An abrupt (within 48-hr) reduction in kidney function defined as an absolute increase in serum creatinine of more than or equal to 0.3 mg/dl, an increase in serum creatinine of more than or equal to 1.5 fold from the value preceding the abnormal value, or reduction in urine output (oliguria of less than 0.5 ml/kg per hour for >6-hr).

Enrollment

All children with features of shock as per standard definitions will be screened for eligibility. Of these, children who require at least one fluid bolus of 20 ml/kg will be enrolled. The eligible participants would be enrolled after obtaining informed consent from one of the parents.

Randomization

Once enrolled, the participants would be randomized into 2 groups. 'MES' or 'study group' will receive the balanced fluids and 'saline' or 'control group' will receive 0.9% saline. Process of randomization will be done by an investigator who will have no further role in collecting the baseline variables, applying intervention or analysis of outcome(s). Block randomization will be done in varying block sizes of 2 to 8. The random number table generated from computer software would be used for this purpose.

Sample size estimation

The investigators calculated that a sample size of 354 patients in each group (708 total) would be required to detect an absolute reduction in incidence of AKI from 25% (current incidence in children with shock in the unit) to 15% assuming a two-sided α level of 0.05 and a statistical power of 90%. The sample size was calculated using Stata 11. The investigators expect the required sample size to be collected within 3 years period in the three centers.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 month to ≤ 15 years with features of septic shock - defined as children who have a suspected infection manifested by hypothermia or hyperthermia and have at least two clinical signs of decreased perfusion with or without hypotension

Exclusion Criteria:

* Children receiving fluid boluses before enrollment
* Children with cardiogenic shock
* Known patient with chronic kidney disease with baseline deranged renal function (eGFR < 90 ml/1.73 m2/min)
* Severe malnutrition
* Children whose parents refuse to give an informed consent

Ages: 2 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 708 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
New or progressive acute kidney injury defined as increase in serum creatinine by > 0.3mg/dL within 48 hours or to 1.5 times baseline or more within the last 7 days or urine output less than 0.5 mL/kg/h for 6 hours | From the time of randomization/intervention to 7 days of admission
  Incidence of new or progressive AKI in first 7 days after randomization/ intervention

SECONDARY OUTCOMES:
Proportion of patients with serum chloride levels > 108 meq/L at admission, 6, 24, 48 and 72 hours | At 6, 24, 48 and 72 hours after randomization
  Incidence of hyperchloremia
Number of fluid boluses received in the first 6 hours after randomization | From the time of randomization to 6 hours
  Total number of fluid boluses received in the first 6 hours after randomization/intervention
Total fluids received in the first 24 hours, 24-48 hours and 48-72hrs in ml/kg after randomization | From the time of randomization to 72 hours
  Total fluids received in first 24 hours, 24-48 hours and 48-72 hours
Mortality (serious adverse event) | From the time of randomization till death or discharge from ICU, whichever came first assessed upto 100 days
  Death during ICU course
Time to resolution of AKI | From the time of onset of AKI after randomization till death or discharge from hospital, whichever came first assessed upto 100 days
  Time taken for resolution of AKI
SOFA scores at 24 and 48 hours after randomization | At 24 and 48 hours after randomization
  Comparison of SOFA scores in both groups at 24 hours and 48 hours after randomization
PELOD scores at 24 and 48 hours after randomization | At 24 and 48 hours after randomization
  Comparison of PELOD scores in both groups at 24 hours and 48 hours after randomization
Incidence of metabolic acidosis at 6, 24, 48 and 72 hours after randomization | At admission and at 6, 24, 48 and 72 hours after randomization
  Comparison of number of children in both groups with acidosis at 6, 24, 48 and 72 hours after randomization

OTHER OUTCOMES:
Safety outcome 1 | From the time of randomization/intervention to 7 days of admission
  New or progressive AKI requiring dialysis (serious adverse event)
Safety outcome 2 | From the time of randomization/intervention to mortality
  IN-ICU mortality in patients with AKI (serious adverse event)
Safety outcome 3 | From the time of initiating the bolus to its completion
  Infusion related adverse events- fever, rash, extravasation, hypervolemia/fluid overload

CONTACTS AND LOCATIONS:
Overall Officials: Jhuma Sankar, MD Ped, Principal Investigator — All India Institute of Medical Sciences; Sushil K Kabra, MD Ped, Study Chair — All India Institute of Medical Sciences; Rakesh Lodha, MD Ped, Study Director — All India Institute of Medical Sciences
Locations (4):
- India (4):
  - St Johns Medical College and Hospital, Bengaluru, Karnataka
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - PGIMER, Chandigarh
  - JIPMER, Puducherry

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared

REFERENCES:
- [Derived] Sankar J, Muralidharan J, Lalitha AV, Rameshkumar R, Pathak M, Das RR, Nadkarni VM, Ismail J, Subramanian M, Nallasamy K, Dev N, Kumar UV, Kumar K, Sharma T, Jaravta K, Thakur N, Aggarwal P, Jat KR, Kabra SK, Lodha R. Multiple Electrolytes Solution Versus Saline as Bolus Fluid for Resuscitation in Pediatric Septic Shock: A Multicenter Randomized Clinical Trial. Crit Care Med. 2023 Nov 1;51(11):1449-1460. doi: 10.1097/CCM.0000000000005952. Epub 2023 Jun 9. PMID 37294145